CLINICAL TRIAL: NCT03272672
Title: Effects of a Valgus Unloader Brace on Medial Femoral Cartilage Changes Following Walking Protocol
Brief Title: Effects of a Valgus Unloader Brace on Medial Femoral Cartilage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 17-0831
Record Dates: First submitted 2017-08-28; First posted 2017-09-05 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded investigator will segment all Ultrasound images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braced (Experimental): Össür Unloading Knee Brace used during walking protocol
  Interventions: Other: Össür Unloading Knee Brace
- Unbraced (No Intervention): Walking protocol without the use of brace

INTERVENTIONS:
Other: Össür Unloading Knee Brace — During the braced walking condition, a valgus unloader brace (Össür Unloader One®, Össur Americas, Orange County, CA) will be fitted by a certified athletic trainer per manufacturer instructions to the dominant limb while the participant is seated with knee flexed to approximately 80°.
  The brace will be maximally adjusted to unload the medial compartment.
  Other Names: Össür Unloader One®
  Arms: Braced

SUMMARY:
The purpose of this study is to determine the effect of a valgus unloader brace condition on the acute change in medial femoral condyle cartilage morphology using Ultrasound following a standardized walking protocol.

DETAILED DESCRIPTION:
Participants will report to an initial screening session during which knee alignment will be determined using a long-lever goniometer. For the assessment of baseline knee alignment, the participant will stand with feet facing forward directly underneath corresponding acromion processes and weight evenly distributed. The first axis will be measured from ASIS to midpoint of the patella and the second axis will be measured from the midpoint of the patella to the tibial tuberosity. The valgus angle will be used to determine eligibility for the study. To be eligible for this study, participants must present with a valgus knee alignment angle of ≥180° on the dominant limb defined as the limb the participant would use to kick a ball. Weight and height measurements will also be measured and used to calculate BMI. Once eligible, participants will determine a self-selected walking speed by walking between 2 sets of infrared timing gates (TF100, TracTronix). Starting approximately 5 steps before the first timing gate, participants will be instructed to walk at a speed described as "comfortable walking over a sidewalk". Each participant will complete 3 trials and the average walking speed will be calculated.

Pre-loading Protocol

Participants will report to the laboratory at the same time of day (±2 hours) for both sessions to account for diurnal variations within the cartilage. Upon arrival, participants will sit on a treatment table in the long-sit position with knees fully extended for 45 mins to allow time for cartilage reformation.

Ultrasonographic Assessment of the Femoral Articular Cartilage While seated with their back up against the wall, participants will flex their knee to 140° measured using a manual goniometer while. A measuring tape will be secured to the length of the table so that the position of the posterior calcaneus can be recorded to allow for consistent positioning across trials 15. A LOGIQe US system (General Electric Co., Fairfield, CT) with a 12MHz linear probe will be used to image both the medial and lateral femoral cartilage. The probe will be placed transversely in line between the medial and lateral femoral condyles just superior to the patella and rotated to maximize reflection off the articular cartilage. A transparent grid will be placed over the US screen to improve reproducibility of the US image. The midpoint of the intercondylar groove will be aligned with the center of the grid.

The level of the cartilage-bone interface at the edge of the image on either side will be recorded in order to ensure consistent positioning across US assessments. Three images will be collected of each knee at each time point. Following each loading condition, the participant will be placed in the same position as the pre-loading US assessment using the tape measure. Three images of the femoral cartilage will be recorded from each knee. All post-walking images will be captured within 5 minutes of the loading protocol.

Ultrasonographic Image Analysis All US images will be analyzed with the ImageJ software (National Institutes of Health, Bethesda, MD). Values for all measurement types will be obtained for each of the three images of the dominant limb at each time point (pre and post-walking) and averaged for statistical analysis.

Cartilage Thickness

Cartilage thickness (in millimeters) will be determined at the most inferior point of the intercondylar groove, the midpoint of the medial condyle, and the midpoint of the lateral condyle by drawing a line from the cartilage-bone interface to the synovial space-cartilage interface.

Cartilage Area The femoral cartilage will be divided into medial and lateral sections by identifying the midline at the most inferior point of the intercondylar groove. Each section of the cartilage will be outlined with a polygon function (Figure 1). The area (in square millimeters) of each section will be measured.

Average Cartilage Thickness The area (in square millimeters) of each section as determined in the cartilage area measure will then be divided by the length (in millimeters) of the section measured via a segmented line along the cartilage-bone interface (Figure 2). Average cartilage thickness (in millimeters) measures will be determined for the medial and lateral condyles. Values will be obtained for each of the three images per limb at each time point (pre and post-walking) and averaged for statistical analysis.

Cartilage Loading Protocol Immediately following pre-test ultrasound assessments, participants will be transferred from the table to a wheelchair in order to minimize knee loading not related to the walking condition. During the braced walking condition, a valgus unloader brace (Össür Unloader One®, Össur Americas, Orange County, CA) will be fitted by a certified athletic trainer per manufacturer instructions to the dominant limb while the participant is seated with knee flexed to approximately 80°.

The brace will be maximally adjusted to unload the medial compartment. The participant will take 30 steps to adjust to the brace. Adjustments will then be made as needed if the participant determines the fit is uncomfortable or too loose. The participant will take 30 more steps. Any final adjustments can be made at that point. The participant will then be transferred to and from the treadmill via wheelchair to control the amount of cartilage loading.

Control Protocol In the unbraced condition, the participant will repeat the brace protocol except that the participant will not be fitted with an unloader brace while seated. The participant will take 60 steps to keep the number of steps consistent across trials before being transferred to the treadmill. The participant will remain unbraced for the entire trial.

Loading Protocol Participants will maintain the self-selected walking speed for 5000 steps on a treadmill (4Front, WOODWAY, Waukesha, WI). Self-selected speed will be kept the same across both conditions. Participant will walk for 1 minute to adjust to treadmill. Steps will then be counted for 1 minute, and the time necessary to complete 5000 steps will be calculated (5000 divided by number of steps per minute).

ELIGIBILITY:
Inclusion Criteria:

* Uninjured participants. There will be no exclusion based on race, gender or ethnicity.

Exclusion Criteria:

* congenital or degenerative joint condition, orthopedic implants, current joint pain (quantified as less than 2 on a 10cm visual analog scale),
* cartilage injury of any joint, lower extremity fracture, or upper extremity fracture within the last year.
* any major ligamentous or cartilage injury of the knee or hip joints, or reported of cartilage injury at the ankle.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Pre walking - Thickness (mm) of the Medial Femoral Articular Cartilage as measured by ultrasound | Prior to the walking protocol
  Thickness of the articular cartilage on the Medial Femoral condyle will be measured in millimeters
Post walking - Thickness (mm) of the Medial Femoral Articular Cartilage as measured by ultrasound | Immediately following the walking protocol (the post-test will be finished within approximately 5 minutes of concluding the walking protocol)
  Thickness of the articular cartilage on the Medial Femoral condyle will be measured in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Valentine, Principal Investigator — University of North Carolina, Chapel Hill; Brian Pietrosimone, PhD, Study Chair — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided